CLINICAL TRIAL: NCT03114488
Title: Modulating Human Cortical Plasticity With Transcranial Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1703M09401
Record Dates: First submitted 2017-03-22; First posted 2017-04-14 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Anodal Stimulation (Experimental)
  Interventions: Device: tDCS
- Sham Stimulation (Sham Comparator)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Transcranial electrical stimulator

SUMMARY:
Experience dependent plasticity is a fundamental property of the brain. It allows neural systems to adapt in response to environmental input and subserves the vital functions of learning and memory. Deficits in plasticity are also thought play a causal role in the pathophysiology of several psychiatric disorders, specifically schizophrenia (SZ). Treatments that can probe or even enhance plasticity have potential to be of great clinical and research value. Non-invasive neuromodulation via transcranial direct current stimulation (tDCS) is a promising method for modulating neural plasticity. tDCS delivers low-intensity direct current to cortical areas, thereby facilitating or inhibiting neural activity in a polarity specific manner. Due to its low cost and safety, tDCS has been employed in a wide variety of studies, but much remains unknown regarding its mechanism of action in humans. Experiments carried out in animal and tissue models indicate that tDCS modulates synaptic plasticity mechanisms of long term potentiation and depression (LTP/D), however, these findings have never been translated to human subjects, limiting the practical utility of the research. Recently developed electroencephalographic (EEG) based measures now allow the interrogation of synaptic plasticity non-invasively in humans, making it possible to explore the effects of tDCS on human brain plasticity.

DETAILED DESCRIPTION:
Experience dependent plasticity is a fundamental property of the brain. It allows neural systems to adapt in response to environmental input and subserves the vital functions of learning and memory. Deficits in plasticity are thought play a causal role in the pathophysiology of several psychiatric disorders, including schizophrenia (SZ). Treatments that can probe or even enhance plasticity have potential to be of great clinical value. Non-invasive neuromodulation via transcranial direct current stimulation (tDCS) is a promising method for modulating neural plasticity. tDCS delivers low-intensity direct current to cortical areas, thereby facilitating or inhibiting neural activity in a polarity specific manner. Its positive effects in a wide range of neurological conditions, as well as its tolerability and low cost, have catalyzed the use of tDCS as a clinical tool. However, issues regarding efficacy and variability of outcomes continue to limit the clinical potential of this promising intervention. Investigation of the physiological mechanisms that subserve tDCS effects in humans is needed to inform treatment protocols and enhance efficacy.

Studies in tissue models have revealed that direct current application alters membrane polarization and modulates long-term potentiation and depression (LTP/D), key mechanisms of synaptic plasticity. In Vivo application of tDCS has been shown to modulate LTP and learning in the rat hippocampus and motor cortex. This modulation was shown to be, persistent, input-specific, and N-methyl-D-aspartate receptor (NMDAR) dependent. These works demonstrate the utility of tDCS in modifying plasticity and learning. Given the limitations placed on invasive procedures, investigating the effects of tDCS on plasticity in the human brain has proved to be much more challenging, limiting the translation and thus the practical utility of the basic research. Utilizing modern, non-invasive methods to probe plasticity in humans has the potential to bridge this translational gap.

Recently developed techniques utilizing electroencephalography (EEG) now enable the non-invasive interrogation of plasticity in the human cortex. Clapp et al., (2005) demonstrated the feasibility of inducing LTP in the cortex by rapid presentation of visual or auditory stimuli, observable as changes in sensory evoked potentials recorded from the scalp. This paradigm, termed stimulus specific plasticity (SSP), is a direct parallel to the high frequency electrical stimulation protocols used to elicit LTP in tissue preparations and satisfies the cardinal features of Hebbian plasticity. Thus sensory-induced plasticity is a useful measure of cortical plasticity that is readily translatable from animals to humans. Further, several studies have used SSP to reveal plasticity deficits in SZ and bipolar disorder, demonstrating the clinical relevance of this assay. In addition, because SSP is a functionally relevant manifestation of LTP, it enables assessment of the efficacy of interventions that target plasticity mechanisms, making it the perfect tool to use for evaluating tDCS effects.

The premise of this proposal is based on prior findings demonstrating the modulatory effect of tDCS on synaptic plasticity in animal and tissue models. Due to methodological limitations, very little work has been done to translate these findings to humans. Because the direct effects of tDCS on plasticity in the humans remains uninvestigated, the overarching goal of this proposal is to assess the in vivo efficacy of tDCS in modulating synaptic plasticity in the auditory cortex of the human brain. To this end, the researchers will conduct a study featuring simultaneous tDCS and EEG recording in a both healthy participants and SZ patients. The two separate cohorts will be randomized into either three or two treatment arms (cathodal, anodal, sham - healthy participants / Anodal and Sham - SZ patients). All subjects will undergo EEG recording during presentation of auditory tones to establish baseline auditory evoked potentials (AEP). LTP will be induced by a high frequency presentation (sensory tetanus) of that same tone for 5 min. Stimulation will begin 10 min prior to the LTP induction and will stop at the end the 5 min period. Post-tetanus EEG recordings of AEP's will be compared to baseline AEP's to analyze the impact of tDCS on neural plasticity.

Specific Aim 1: Evaluate the effects of Anodal tDCS vs. Cathodal tDCS vs. Sham on induction of LTP in a healthy population: Significant findings demonstrate that anodal tDCS impacts neuronal function by enhancing LTP induction. Based on these findings in animal and tissue models, it is expected that anodal tDCS will lead to a greater facilitation of LTP than cathodal or sham stimulation Specific Aim 2: Evaluate the efficacy of Anodal tDCS in enhancing induction of LTP in a population of SZ Patients: SZ patients show deficient capacity to support LTP in the auditory cortex. Effect of tDCS are putatively emergent from modulation of NMDAR dependent plasticity mechanisms. Using the SSP paradigm the study will evaluate the efficacy of tDCS in modulating LTP measures. Based on mechanistic work in animals demonstrating the NMDAR dependent action of tDCS, it is expected that anodal tDCS will enhance the induction of LTP compared to sham.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* No psychiatric medication prescription
* No clinically significant head injury or neurological disease
* No dependence in the past 6 month or no substance abuse in the past month
* Sufficient spoken english to understand testing procedures
* Ability to give informed consent

Exclusion Criteria:

* History of transcranial electrical stimulation (tES) or other cortical energy exposure in the past 12 months; including
* participation in any neuromodulation studies
* History of seizures or epilepsy
* History of metallic cranial plates, screws, or implanted device
* History of craniotomy
* History of eczema on the scalp
* History of traumatic brain injury
* History of mental illness (Healthy group)
* Diagnosis of bipolar disorder
* Diagnosis of major depression
* Unable to give informed consent
* Hairstyle that is braided in cornrows or in dreadlocks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kelvin O. Lim, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS First, Then Sham: Participants randomized to active tDCS first, then the sham treatment
- Sham tDCS First, Then Active: Participants randomized to sham tDCS first, then the active treatment
Period: Time Period 1
Arm/Group | Active tDCS First, Then Sham | Sham tDCS First, Then Active
Started | 19 | 22
Completed | 19 | 22
Not Completed | 0 | 0
Period: Time Period 2
Arm/Group | Active tDCS First, Then Sham | Sham tDCS First, Then Active
Started | 19 | 22
Completed | 18 | 19
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Crossover Design: All participants are included in baseline analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Amplitude of N100 Component of the Auditory Evoked Potential
Description: The amplitude of the N100 component will be averaged across individuals in each group. Grand averages from the two groups will be compared. Outcome is reported as the change from baseline to post-treatment (approximately 1 hour).
Time Frame: approximately 1 hour
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- Anodal Stimulation - Time Period 1: Change from baseline to post-treatment of Amplitude of N100 component of the Auditory Evoked potential
  Crossover design, experimental stimulation arm - time period 1
- Sham Stimulation - Time Period 1: Change from baseline to post-treatment of Amplitude of N100 component of the Auditory Evoked potential
  Crossover design, sham stimulation arm - time period 1
- Anodal Stimulation - Time Period 2: Change from baseline to post-treatment of Amplitude of N100 component of the Auditory Evoked potential
  Crossover design, experimental stimulation arm - time period 2
- Sham Stimulation - Time Period 2: Change from baseline to post-treatment of Amplitude of N100 component of the Auditory Evoked potential
  Crossover design, sham stimulation arm - time period 2
Arm/Group | Anodal Stimulation - Time Period 1 | Sham Stimulation - Time Period 1 | Anodal Stimulation - Time Period 2 | Sham Stimulation - Time Period 2
Number analyzed (Participants) | 19 | 22 | 18 | 19
microvolts | -1.1 (1.18) | -0.35 (0.543) | -0.77 (1.22) | -0.33 (0.661)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Anodal Stimulation - Time Period 1 | Sham Stimulation - Time Period 1 | Anodal Stimulation - Time Period 2 | Sham Stimulation - Time Period 2
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22 | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03114488/Prot_SAP_000.pdf